CLINICAL TRIAL: NCT03614780
Title: Environmental Exposures Across Urban and Rural Communities in the Deep South
Brief Title: Pre Post Evaluation of Temperature, Steps, and Glucose With Additional Time Spent Outdoors in an Urban and Rural Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: University of Alabama at Birmingham (Other); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Julia Gohlke, Associate Professor, Virginia Polytechnic Institute and State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-761; R01ES023029 (NIH)
Record Dates: First submitted 2018-07-27; First posted 2018-08-03 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Temperature; Exercise; Diabetes Mellitus, Type 2
Keywords: rurality
MeSH Terms: conditions — Motor Activity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 30 additional minutes outdoors (Experimental): Participants were asked to go about their normal activities during the first 2 baseline days of participation. Participants were asked to spend an additional 30 minutes outdoors per day for the next 5 days of participation.
  Interventions: Behavioral: 30 minutes outdoors

INTERVENTIONS:
Behavioral: 30 minutes outdoors — Participants were asked to add an additional 30 minutes of time spent outdoors during the last 5 days of participation

SUMMARY:
This research was designed with partners to determine differences in temperature exposures in urban and rural communities in Alabama. The investigators hypothesized that significant differences in temperature exposure exist between urban and rural settings. Time spent outdoors has been previously positively associated with greater physical activity. Built environment components in urban versus rural environments and ambient temperatures experienced during the summer may pose barriers to time spent outdoors. Persons with Type II Diabetes Mellitus may find it more difficult to overcome temperature barriers due to reduced thermoregulation capacity. This analysis will result in a more precise picture of temperature exposure as well as behavioral factors that may mediate exposure.

DETAILED DESCRIPTION:
The investigators gathered individual-level temperature exposure data by asking 180 female participants to wear a small thermometer on their shoe for 7 days. Ninety participants were recruited from Birmingham AL (urban) and 90 from rural West Central Alabama. The first two days participants were asked to go about their normal daily activities. During the next 5 days of participation, participants were asked to add an additional 30 minutes of time spent outdoors. As a secondary outcome, steps were measured via pedometers worn by participants. A subgroup of participants with self-reported doctor diagnosed Type II Diabetes also recorded their fasting glucose each morning of participation.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 19 to 65, willing to wear a small thermometer on shoe and pedometer on waist for one week.

Exclusion Criteria:

* Medical condition that limits the amount of time able to be spent outdoors.

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
temperature | 7 days
  participants wore a small thermometer on their shoe that recorded temperature in 5 minute intervals for the duration of participation

SECONDARY OUTCOMES:
steps | 7 days
  participants wore a pedometer and recorded steps daily
fasting glucose | 7 days
  Participants (N=46) that self reported diagnosed T2DM and measured daily fasting glucose were asked to log their fasting glucose level each morning.

CONTACTS AND LOCATIONS:
Overall Officials: Julia M Gohlke, PhD, Principal Investigator — Virginia Polytechnic Institution and State University
Locations (1):
- Center for the Study of Community Health, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No